CLINICAL TRIAL: NCT03013413
Title: Evaluation of the Aixplorer Ultrasound System for Evaluation of the Prostate
Brief Title: Ultrasound-Based Imaging Using the Aixplorer System in Diagnosing Prostate Cancer in Patients Undergoing Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11D.349; JT 1614 (Other: JeffTrial Number)
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic (elastography imaging using the Aixplorer system) (Experimental): Patients undergo ultrasound-based elastography imaging using the Aixplorer system followed by standard of care ultrasound-guided prostate biopsy over approximately 25 minutes.
  Interventions: Procedure: Shear Wave Elastography; Procedure: Ultrasound Elasticity Imaging; Procedure: Ultrasound-Guided Prostate Biopsy

INTERVENTIONS:
Procedure: Shear Wave Elastography — Undergo ultrasound-based elastography imaging using the Aixplorer system
  Other Names: Transient Elastography
Procedure: Ultrasound Elasticity Imaging — Undergo ultrasound-based elastography imaging using the Aixplorer system
Procedure: Ultrasound-Guided Prostate Biopsy — Undergo standard of care ultrasound-guided prostate biopsy

SUMMARY:
This clinical trial studies an ultrasound-based imaging procedure called elastography using the Aixplorer system in diagnosing prostate cancer in patients undergoing biopsy. Ultrasound is a non-invasive imaging technique that uses high-frequency sound waves to produce images of internal structures. Elastography uses ultrasound imaging techniques to examine the stiffness or elasticity of a tissue and may enhance the detection of prostate cancer. It is not yet known whether elastography imaging using the Aixplorer system works better than standard ultrasound imaging in detecting prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the detection of prostate cancer with elastography using the Aixplorer scanner.

SECONDARY OBJECTIVES:

I. To obtain quantitative data on the elastic properties of normal and malignant tissue in the prostate of patients referred for ultrasound guided biopsy.

II. To compare the Gleason grade of prostate cancers detected with elastography to the Gleason grade of tumors detected by conventional systematic biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Be scheduled for a clinically indicated biopsy of the prostate
* Agree to an ultrasound examination using the Aixplorer system
* Sign an institutional review board (IRB) approved informed consent prior to any study procedures

Exclusion Criteria:

• Recent prostate biopsy within 90 days

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2011-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Frequency of diagnosis of prostate cancer using elastography using the Aixplorer scanner | At the time of prostate biopsy
  Will focus on comparing the frequency of diagnosis of prostate cancer between conventional systematic biopsy and targeted biopsy based upon abnormalities in gray scale imaging, Doppler imaging, and elastography. The main parameter of interest will be the ratio of the detection frequency with targeted biopsy versus that with systematic biopsy. The analyses will be based on methods for matched data in cohort studies and will use the appropriate estimate and variance for the relative risk.

SECONDARY OUTCOMES:
Gleason scores of the cores detected with targeted biopsy versus those of the cores of systematic biopsy | At the time of prostate biopsy
  Analyses will be carried out via the Generalized Estimating Equations methods to account for clustering within patient (multiple cores per patient).

CONTACTS AND LOCATIONS:
Overall Officials: Ethan Halpern, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Sidney Kimmel Cancer Center — http://www.kimmelcancercenter.org
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/